CLINICAL TRIAL: NCT01944683
Title: Phase 1b Study of Pharmacokinetic Interaction, Evaluating the Effect of a Single IV Infusion of GGF2 or Placebo on Midazolam Pharmacokinetics in Patients With Heart Failure
Brief Title: A Double-Blind Pharmacokinetic Interaction Study Evaluating the Effect of a Single IV Infusion of GGF2 or Placebo on Midazolam Pharmacokinetics in Patients With Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GGF2-CV-1007
Record Dates: First submitted 2013-09-11; First posted 2013-09-18 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GGF2 (Experimental): Patients will be randomized to receive GGF2 or Placebo and on study day 3 administered a single IV infusion.
  Each patient will receive 5 oral doses of Midazolam syrup on study day 1 and days 4 through 7 respectively.
  Interventions: Drug: GGF2; Drug: Midazolam
- Placebo (Placebo Comparator): Patients will be randomized to receive GGF2 or Placebo and on study day 3 administered a single IV infusion.
  Each patient will receive 5 oral doses of Midazolam syrup on study day 1 and days 4 through 7 respectively.
  Interventions: Other: Placebo; Drug: Midazolam

INTERVENTIONS:
Other: Placebo
  Arms: Placebo
Drug: GGF2
  Arms: GGF2
Drug: Midazolam

SUMMARY:
The study will examine midazolam pharmacokinetics following single dose administration of 3 planned dose levels of GGF2 .

DETAILED DESCRIPTION:
This drug-drug interaction (DDI) study evaluates the potential effect of intravenously administered GGF2 on the elimination kinetics of midazolam.

ELIGIBILITY:
Inclusion Criteria:

* If female, must be at least 2 years post-menopausal or have bilateral oophorectomy, hysterectomy or documented sterility
* If male, must have documented sterility (by verbal report or previous vasectomy), or if non-sterile, must agree to use barrier contraception for the entire duration of the trial and until 3 months after the last dose of investigational product. Must also agree not to donate sperm during the study and up to 3 months after the last dose of investigational product
* Stable coronary disease without unstable angina or acute coronary syndrome in the last 6 months
* All cardiac medications, specifically beta-blockers, renin-angiotensin system inhibitors, aldosterone antagonists, hydralazine and nitrates are at a stable dose (at least 4 weeks) prior to Day 1

Exclusion Criteria:

* Any previous exposure to GGF2 or other neuregulins
* Initiation or change of a prescription medication within the 2 weeks prior to Day 1, and/or concomitant medication regimen is expected to change during the course of the study
* Known allergic reaction to midazolam, or any of the components of midazolam syrup (including cherry flavoring), or components of GGF2 diluent
* Known specific hepatic disease; total bilirubin >2 mg/dL, AST > 100 IU
* History of hepatic impairment (hepatitis B and C)
* Type I Diabetes
* Documented stroke or transient ischemic attack (TIA) within 2 months of study enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-09; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of GGF2 IV infusion in patients with heart failure assessed by review of Treatment Emergent Adverse Events (TEAE) | 90 days (± 3 days)
Pharmacokinetic (PK) parameter Area Under the Curve (AUC) of a single dose of midazolam when administered prior to and following a single IV infusion of GGF2 or Placebo | Day 1 to Day 7

SECONDARY OUTCOMES:
Change from baseline of 2D-Echocardiogram (2D-ECHO) or ECHO with contrast | Visit 1 (day-14 to day-1) and visits 2-5 (day 8 through day 90 ± 3 days)
Change from baseline of the Six-Minute Walk Test (6MWT) | Visit 1 (day-14 to day-1) and visits 3-5 (day 14 through day 90 ± 3 days)
Change from baseline of metabolic testing measuring maximum capacity of body to transport and use oxygen during incremental exercise (VCO2 and VO2 max) | Visit 1 (day-14 to day-1) and visits 3-5 (day 14 through day 90 ± 3 days)
Change from baseline of the M.D. Anderson Symptom Inventory (MDASI) score | Visit 1 (day-14 to day-1) and visits 3-5 (day 14 through day 90 ± 3 days)
  MDASI is a questionnaire asking patients about the severity of their heart disease symptoms and impact of the symptoms on daily functioning during the past 24 hours.
  Scale ranges from 0 (sympton has not been present) to 10 (the symptom was as bad as you can imagine it could be).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Eisen, MD, Study Director — Acorda Therapeutics
Locations (8):
- United States (8):
  - UCSD Medical Center, La Jolla, California
  - Orange County Research Center, Tustin, California
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Duke Clinical Research Unit, Durham, North Carolina
  - New Orleans Center for Clinical Research (NOCCR), Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia